CLINICAL TRIAL: NCT06867120
Title: Bowel Sound in Predicting the Severity of Acute Pancreatitis: Protocol of a Prospective, Multi-center Study
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Beijing Sixth Hospital (Unknown); Beijing Longfu Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2022-PUMCH-B-023
Record Dates: First submitted 2025-01-25; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-01

CONDITIONS: Acute Pancreatitis (AP); Severe Acute Pancreatitis
Keywords: bowel sound; acute pancreatitis; intestinal function; prediction
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational Cohort

SUMMARY:
Introduction: Acute pancreatitis (AP) is a common condition, with 20% of cases progressing to severe acute pancreatitis (SAP), which is associated with a poor prognosis. Early identification of patients likely to progress to SAP is crucial for timely intervention. This study aims to use bowel sound monitoring to predict early progression to SAP in AP patients.

Methods and analysis: This study is a prospective, multi-center prognostic study . Investigators will consecutively recruit newly diagnosed acute pancreatitis (AP) patients at emergency departments across three centers from December 2023. Upon enrollment, each patient will undergo continuous bowel sound monitoring for at least 48 hours using standardized equipment and procedures. The primary outcome is the occurrence of SAP during hospitalization. Collected bowel sound data will be analyzed by an unsupervised automated algorithm to estimate a bowel sound activity index, which serves as the main diagnostic indicator for SAP. This process will be fully blinded to patients' SAP status. Investigators will calculate the ROC curve and area under the curve (AUC) for the bowel sound activity index's ability to diagnose SAP. Additionally, this study will perform exploratory analyses on differences in gut microbiota and serum intestinal permeability markers (diamine oxidase, D-lactic acid, and bacterial endotoxin) between patients with and without SAP. Investigators will also assess whether bowel sound monitoring can reflect these inter-group differences.

Strengths and limitations of the study:

1. Our research aims to monitor bowel sounds in real-time and dynamically, providing an objective tool for monitoring intestinal activity in AP patients.
2. Our research might offer an objective tool to evaluate bowel sounds, aiding in assessing AP patients' intestinal function and complementing existing score systems like the modified Marshall score.
3. By detecting bowel sounds in the early stage of AP, investigators could better monitor intestinal function, which might aid in predicting the prognosis of AP patients.
4. Our monitoring system's main limitation is its difficulty in pinpointing bowel sound changes in specific intestinal segments due to its detection across the entire abdomen.

ELIGIBILITY:
Inclusion criteria:

1. Aged between 18 and 85 years old.
2. Meet the diagnostic criteria for AP, at least two of the following three: (a) characteristic abdominal pain; (b) serum amylase and lipase levels are greater than three times the upper limit of normal; (c) abdominal images with typical manifestations of AP.
3. AP patients within 48 hours of onset.
4. The patient or family members understand the study protocol and sign the informed consent form.

Exclusion criteria:

The patients who fulfill any of the following criteria will be excluded:

1. Patients with serious conditions requiring surgery and abdominal lavage.
2. Pregnant women.
3. The patients with muscle and nerve disorders, chronic pancreatitis, inflammatory bowel disease, cancer, and irritable bowel syndrome.
4. The patients with severe digestive, respiratory, cardiovascular, hematological, endocrine, psychiatric, and infectious diseases.
5. The patients have a history of abdominal surgery (except appendectomy or cholecystectomy).
6. Allergic to silicone, polycarbonate materials or medical plaster. The intake of antibiotic, probiotics, and Chinese herbal medicine will be recorded before the collection of the swabs and will not be considered as exclusion criteria.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study included AP patients admitted to the outpatient/emergency and inpatient wards of Peking Union Medical College Hospital, Beijing Sixth Hospital, and Beijing Longfu Hospital from December 2023 to December 2026.
Sampling Method: Non-Probability Sample
Enrollment: 352 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with severe acute pancreatitis (SAP) during hospitalization within 7 days after enrollment. | Within 7 days after enrollment.
  SAP was defined as AP patients with persistent organ failure according to the revised Atlanta classification.

SECONDARY OUTCOMES:
Number of participants with in-hospital mortality. | Within 30 days after enrollment.
  Number of participants who died during hospitalization.
Number of participants with 30-day mortality. | Within 30 days after enrollment.
  Number of participants who died within 30 days after enrollment.
Length of hospital stay. | Within 30 days after enrollment.
  The number of days participants stayed in the hospital.
Number of participants with organ failure. | Within 30 days after enrollment.
  Number of participants who developed organ failure.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No